CLINICAL TRIAL: NCT05608252
Title: A Single Arm Phase 1/2 Trial of Abemaciclib + VS-6766 + Fulvestrant in Metastatic HR+/HER2- Breast Cancer
Brief Title: VS-6766+Abema+Fulv in Met HR+/HER- BC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adrienne G. Waks (Other)
Collaborators: Verastem, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Adrienne G. Waks, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-490
Record Dates: First submitted 2022-10-27; First posted 2022-11-08 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Hormone Receptor-positive Breast Cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer
Keywords: Breast Cancer; Hormone Receptor-positive Breast Cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): During 28 day/4 week study cycle, participants will receive:
  * VS-6766 2x weekly for 3 out of the 4 week cycle
  * Abemaciclib 2x daily
  * Fulvestrant on day 1 of each study cycle (and day 15 of cycle 1 only)
  Interventions: Drug: VS-6766; Drug: Abemaciclib; Drug: Fulvestrant
- Phase 2 Dose Expansion (Experimental): Participants will receive VS-6766 with abemaciclib and fulvestrant at the recommended phase II doses determined in the phase I portion of the study.
  Interventions: Drug: VS-6766; Drug: Abemaciclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: VS-6766 — Taken Orally
Drug: Abemaciclib — Taken Orally
  Other Names: Verzenio
Drug: Fulvestrant — Administered by intramuscular injection
  Other Names: Faslodex

SUMMARY:
This research is being done to evaluate the safety and effectiveness of a drug currently known as VS-6766 in combination with the drugs abemaciclib and fulvestrant in HR+/HER2-negative breast cancer.

The names of the study drugs involved in this study are:

* VS-6766
* Abemaciclib
* Fulvestrant

DETAILED DESCRIPTION:
This is single-arm open-label phase 1/2 trial assessing the safety and efficacy of the new drug, VS-6766, plus abemaciclib and fulvestrant in treating metastatic hormone receptor-positive and HER2-negative (HR+/HER2-) breast cancer.

VS-6766 is a unique small molecule drug that targets and interrupts a pathway that allows cancer cells to grow.The U.S. Food and Drug Administration (FDA) has not approved VS-6766 as a treatment for any disease. The FDA has approved abemaciclib and fulvestrant as a treatment option for breast cancer.

The study is divided into three study periods: a screening period; a treatment period; and a post-treatment follow-up period. Participants will receive study treatment for as long there are no serious side effects and the disease does not get worse.

It is expected that about 63 people will take part in this research study.

Verastem Oncology, a biopharmaceutical company, is supporting this research study by providing VS-6766 and funding to conduct this trial. Eli Lilly, a pharmaceutical company, is supporting this research study by providing the drug, abemaciclib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed hormone receptor positive (HR+), HER2 negative metastatic or locally recurrent unresectable invasive breast cancer. ER, PR and HER2 measurements should be performed according to institutional guidelines, in a CLIA-approved setting. Cut-off values for positive/negative staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines.
* Participants may have measurable or non-measurable disease according to RECIST v1.1.
* Men and pre- and postmenopausal women are eligible. Ongoing monthly GNRH agonist is required in pre-menopausal women or male participants for at least 4 weeks prior to study entry. If men or pre-menopausal women have not received regular GNRH agonist for at least 4 weeks prior to study entry, these patients will be excluded.
* Participants must have radiological or objective evidence of progression on any CDK 4/6 inhibitor-containing regimen in the metastatic setting, and/or relapse/progression during or within 12 months of completion of any CDK4/6 inhibitor-containing regimen in the adjuvant setting.

  * It is not mandatory to have a CDK4/6 inhibitor-containing regimen as the most recent treatment.
* Participants must have radiological or objective evidence of progression on fulvestrant (as a single agent or as a component of any multi-drug regimen) in the metastatic setting.

  * It is not mandatory to have a fulvestrant-containing regimen as the most recent treatment.
* Prior therapy:

  * No more than two prior chemotherapy regimens in the metastatic setting.
  * For both the phase I and phase II portions of this trial, there is no limit on prior lines of endocrine therapy in the adjuvant or metastatic setting.
* For phase 2 cohort only: Willing to undergo pre- and on-treatment tumor biopsies. Patients are exempt from this requirement if, in the opinion of the investigator, the biopsy procedure would pose a significant risk. Biopsies are optional in the phase 1 cohort.
* ECOG performance status <2.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1.5 x 109/L
  * platelets ≥100,000/μl
  * hemoglobin ≥9 g/dL (If red blood cell transfusion has been administered, hemoglobin must remain stable and ≥9 g/dL without further transfusion for at least 1 week prior to first dose of study therapy).
  * total bilirubin ≤1.5mg/dL (≤3.0mg/dL in patients with known Gilbert syndrome and direct bilirubin within normal limits)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN.
  * Adequate renal function with a creatinine clearance rate of ≥ 50 mL/min as calculated by the Cockcroft-Gault formula.
  * International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 1.5 x ULN in the absence of anticoagulation or therapeutic levels in the presence of anticoagulation.
  * Creatine phosphokinase (CPK) ≤ 2.5 x ULN.
  * Adequate cardiac function with left ventricular ejection fraction ≥ 50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
  * Baseline QTc interval < 480 ms (average of triplicate readings) using Fredericia's QT correction formula. NOTE: This criterion does not apply to patients with a complete or incomplete right or left bundle branch block.
* Adequate recovery from toxicities related to prior systemic treatments, surgery, or radiotherapy to at least Grade 1 by CTCAE v 5.0. Exceptions include alopecia and peripheral neuropathy grade ≤ 2.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of study agents in participants <18 years of age, children are excluded from this study.
* Women of childbearing potential, women who are made postmenopausal through use of GNRH agonists, and men must agree to use adequate contraception for the duration of protocol treatment. Women meeting these criteria will need to use adequate contraception for at least 30 days after the last dose of abemaciclib or VS-6766 and for one year after the last dose of fulvestrant. Men will need to use adequate contraception for 90 days after the last dose of abemaciclib or VS-6766 and for one year after the last dose of fulvestrant. Additionally, males must agree not to donate sperm for the duration of protocol treatment and for at least 90 days after the last dose of protocol therapy. Childbearing potential for this purpose is defined as: those who have not been surgically sterilized and/or have had a menstrual period in the past 12 months. Adequate contraception is defined as one highly effective non-hormonal form of contraception or two effective forms of non-hormonal contraception by the participant and/or partner:

Highly Effective Non-Hormonal Contraception Methods of birth control which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly are considered highly-effective forms of contraception.

The following non-hormonal methods of contraception are acceptable:

* True abstinence when this is in line with the preferred and usual lifestyle of the participant. [Periodic abstinence (e.g., calendar, ovulation, symptothermal post-ovulation methods) and withdrawal are not acceptable methods of contraception].
* Male sterilization (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female participants, the vasectomized male partner should be the sole partner. OR Effective Non-Hormonal Contraception

Alternatively two of the following effective forms of contraception may be used instead:

* Placement of non-hormonal or progesterone-coated intrauterine device (IUD) or intrauterine system (IUS). Consideration should be given to the type of device being used, as there are higher failure rates quoted for certain types, e.g., steel or copper wire.
* Condom with spermicidal foam/gel/film/cream/suppository.
* Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* The use of barrier contraceptives should always be supplemented with the use of spermicide. The following should be noted:
* Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore, the use of additional spermicides does confer additional theoretical contraceptive protection.
* However, spermicides alone are ineffective at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

It should be noted that two forms of effective contraception are required. A double barrier method is acceptable, which is defined as condom and occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

* A female of childbearing potential, as defined above in section 3.1.12, must have a negative serum pregnancy test performed within 7 days of C1D1. A positive urine test must be confirmed by a serum test. Pregnancy testing does not need to be pursued in female participants who are:

  * Age >60 years; or
  * Age <60 years with intact uterus and amenorrhea for 12 consecutive months or more AND estrogen (estradiol) levels within postmenopausal range; or
  * Status post bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation
* Participant must be able to swallow and retain oral medication.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with active brain metastases or with known carcinomatous meningitis. Stable, treated brain metastases are allowed (this includes participants who have documented radiologic stability at least 4 weeks after radiotherapy, and do not require systemic steroids for management of symptoms from CNS metastatic lesions). Any patients with documented brain metastasis not meeting above criteria for stable treated brain metastasis are considered to have active brain metastases.
* Phase I: Participants who have discontinued prior abemaciclib for toxicity, at any dose. Phase II: Participants who have discontinued prior abemaciclib for toxicity, if that toxicity occurred at or above the RP2 dose level for abemaciclib that is incorporated into phase II of this trial.
* Participants who have discontinued prior fulvestrant for toxicity.
* Prior treatment with any MEK inhibitor.
* The subject has received another investigational agent within at least 30 days or 5 half-lives of the first dose of study drug, whichever is longer, or is currently enrolled in any medical device research or other research that is judged by the sponsor to not be scientifically or medically compatible with this study.
* The subject has received a chemotherapy agent or immunotherapy within 21 days of the first dose of study drug.
* The subject has received an endocrine or biologic agent within 14 days of the first dose of study drug.
* The subject has completed radiation within 14 days of registration. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy.
* The subject has had major surgery within 14 days of registration.
* Participants with the following pre-existing ocular pathology are excluded:
* Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
* Patient with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
* Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
* History of rhabdomyolysis or neuromuscular disorders that are associated with elevated CK (eg inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* The patient has an uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure (New York Heart Association Class III or IV), active ischemic heart disease, myocardial infarction within the previous six months, syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), uncontrolled diabetes mellitus, severe obstructive pulmonary disease, or severe chronic liver or renal disease, or sudden cardiac arrest.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are potentially eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years and there is no evidence of disease recurrence for 1 year or more since completion of appropriate therapy: cervical cancer in situ, and non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the overall study PI to determine eligibility.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to VS-6766 (including inactive ingredients mannitol, magnesium stearate, HPMC (hydroxypropylmethylcellulose) shells), abemaciclib, or fulvestrant.
* Known history of testing positive for HIV with history of an AIDS-defining opportunistic infection within the past 12 months, or need to receive combination antiretroviral therapy for HIV that are strong CYP3A4 inhibitors or inducers.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (for example, hepatitis B surface antigen positive). Screening is not required for enrollment. Patients with chronic HBV infection who meet criteria for anti-HBV therapy should be on suppressive antiviral therapy prior to initiation of study therapy. Patients with a history of HCV infection will need to have completed curative antiviral treatment with HCV viral load below the limit of quantification. Patients with untreated HCV may be enrolled if the HCV is stable and if the patient is not at risk for hepatic decompensation. Patients that need to receive antiviral therapy for HBV or HCV that are strong CYP3A4 inhibitors or inducers will be excluded.
* Patients exposed to strong CYP3A4 inhibitors or inducers within 14 days prior to the first dose of study drugs (see Appendix C). Concurrent use of strong CYP3A4 inhibitors (see Appendix C), such as ketoconazole and erythromycin, or inducers (see Appendix C), such as St. John's wort, should be avoided during the study treatment.
* Pregnant women are excluded from this study because effect of combination VS-766, abemaciclib, and fulvestrant on a developing fetus is unknown. Breastfeeding should be discontinued prior to entry onto the study.
* Patients with the inability to swallow oral medications, impaired gastrointestinal absorption due to gastrectomy or other major surgical resection involving the stomach or small bowel, preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea, or other medical issue that would impact absorption of oral medication in the opinion of the investigator.
* Patients with active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), or fungal infection (requiring IV antifungal treatment at time of initiating study treatment), or severe acute respiratory syndrome from coronavirus 2 (SARS-Cov2) infection ≤28 days prior to first dose of study treatment.
* Patients on treatment with warfarin. Individuals on treatment with warfarin must be transitioned to anticoagulation instead with low-molecular-weight heparin or a direct oral anticoagulant prior to first dose of study treatment.
* Any other serious and/or uncontrolled preexisting medical condition(s) (e.g. interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, other cardiac, gastrointestinal, pulmonary, psychiatric, neurological, or genetic conditions, etc.) that in the opinion of the Investigator would place the patient at unacceptably high risk for toxicity and therefore preclude participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Maximum tolerated dose (MTD) | 4 Weeks up to 2 years
  Determine maximum tolerated dose (MTD) of VS-6766 in combination with abemaciclib and fulvestrant using Bayesian Optimal Interval Design
Phase 1 Recommended Phase II Dose (RP2D) | 4 Weeks up to 2 years
  Determine Recommended Phase II Dose (RP2D) of VS-6766 in combination with abemaciclib and fulvestrant using Bayesian Optimal Interval Design
Phase 2 Clinical benefit rate (CBR) | 6 months up to 3 years
  The primary endpoint in phase II is assessment of the clinical benefit rate (CBR; complete response + partial response + stable disease for >/=24 weeks)

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months up to 3 years
  Assess overall response rate (ORR) defined as confirmed complete response or partial response per RECIST 1.1.
Progression-free survival (PFS) | 6 months up to 3 years
  Assess progression-free survival (PFS) defined as as the time from study registration to radiographic or clinical evidence of disease progression or death due to any cause, whichever occurred first. Patients alive without disease progression are censored at the date of last disease evaluation.
Overall survival (OS) | 6 months up to 10 years
  Assess Overall survival (OS) defined as time from randomization (or registration) to death due to any cause, or censored at date last known alive.
Treatment Related Adverse Events | 1 week up to 3 years
  Assess safety through number of Treatment Related Adverse Events per CTCAE v5.0
Phase I Cmax of VS-6766 | 16 days
  In Phase 1 define the maximum concentration of drug VS-6766
Phase I Cmax of abemaciclib | 16 days
  In Phase 1 define the maximum concentration of drug abemaciclib
Phase I AUC(0-384) of VS-6766 | 16 days
  In Phase 1 define the area under the curve (AUC) from 0-384 hours of VS-6766
Phase I AUC(0-384) of abemaciclib | 16 days
  In Phase 1 define the area under the curve (AUC) from 0-384 hours of abemaciclib

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne G Waks, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institite, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu